CLINICAL TRIAL: NCT04554641
Title: The Effect of a Multi-strain Live Bacteria Supplement on the Gut Microbiota Composition of Healthy Adults: an Open Label Trial
Brief Title: Effect of a Multi Strain Probiotic on the Gut Microbiota
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Functional Gut Clinic (Other)
Collaborators: ADM Protexin (Industry)
Responsible Party: Principal Investigator, Dr Anthony Hobson, Consultant Clinical Scientist, The Functional Gut Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: FGC-19-003
Record Dates: First submitted 2020-09-04; First posted 2020-09-18 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Microbial Colonization
Keywords: Probiotics; Microbiome; Gastrointestinal
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BioKult Advanced (Experimental): This is a single arm study, all participants will take Bio-kult Advanced for 56 days (+/- 2days). Participants will be required to take 4 capsules daily.
  Interventions: Other: Fasted breath samples; Other: Daily Diary; Other: Stool sample

INTERVENTIONS:
Other: Fasted breath samples — Participants will provide fasted breath samples pre and post Bio-Kult Advanced.
Other: Daily Diary — Monitoring stool form, consistency and frequency on a daily basis.
Other: Stool sample — Participants will provide stool sample pre and post Bio-kult Advanced.

SUMMARY:
Over recent years there has been a lot of research looking at how the bacteria in our gut affect our health. Changes to gut bacteria has been linked to several diseases. Taking specific live bacteria supplements (sometimes known as 'probiotics'), to change the balance of our gut bacteria to result in a health benefit have been trialled as a treatment option for many diseases in recent years.

Bio-Kult Advanced is a live bacteria Food supplement that contains 14 different bacteria cultures. The effect of Bio-Kult Advanced on gut bacteria is unknown, therefore, the aim

DETAILED DESCRIPTION:
There is rapidly growing interest in the involvement of the microbiome in health. Imbalance in human gut microbiota, 'dysbiosis', has been linked to several diseases. Manipulation of the microbiome, using specific strains of live micro-organisms, that confer a health benefit on the host (probiotics), have therefore become an exploratory treatment option in microbiome-associated diseases in recent years. Numerous studies have shown selected strains of bacteria to show statistically significant and clinically relevant improvement in symptoms, in a number of diseases, including but not limited to infantile colic and atopic dermatitis.

Bio-Kult Advanced (BKA) is a 14 strain live bacteria supplement containing a Minimum 2 billion live microorganisms per capsule (2x109 CFU/capsule), equivalent to 10 billion live microorganisms per gram (1x1010 CFU/gram). A randomised controlled trial of Bio-Kult Advanced in the management of diarrhoea predominant IBS demonstrated significant improvement in gastrointestinal (GI) symptoms and was well tolerated by participants. Another randomised controlled trial of Bio-Kult Advanced, in participants with episodic and chronic migraine sufferers, demonstrated significant improvement in frequency and severity of migraines compared to placebo. This clinical effectiveness across various conditions, suggest that bacterial strains in Bio-Kult could have an effect on the gastrointestinal flora, however data has yet to be collected that explores the effect of Bio-Kult on the microbiome. The aim of this study is to therefore investigate the effect of Bio-Kult Advanced, on the composition of the gut microbiota in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Adult males and females (50:50) between 18 to 40 years old
* No significant medical diagnosis (healthy individuals)
* Not on regular prescription medicines
* No selective/restricted diets (e.g. vegan, low FODMAP)
* Body Mass Index of 18.50-29.99 kg/m2
* Participant able to understand the participant information sheet in English and provide informed consent

Exclusion Criteria:

* Diagnosis of any medical condition, except for visual impairment and other conditions to clinicians discretion
* Prior abdominal surgery (e.g. appendectomy, bariatric surgery )
* Migraine as based on migraine definition by ICHD 2019:

  * A minimum of five attacks (in absolute terms) fulfilling criteria:

    * Duration 4 - 72 hours
    * At least two of the following:
* unilateral location
* pulsating character
* moderate or severe pain intensity
* aggravation by routine physical activity
* Presence of nausea/vomiting OR photophobia/phonophobia during headache
* Ongoing therapy with medication known to affect the gut microbiome:

  * Antibiotics used in the last 8 weeks
  * Proton pump inhibitors used in the last 8 weeks
  * Antidepressants in the last 8 weeks
  * Regular use of laxatives or anti-diarrheal medications
* Alcohol consumption >14 units per week
* Pregnancy or breastfeeding
* Vegan and other selective diets, use of diet replacements (e.g. Huel)
* Regular consumption of probiotics, prebiotics, fibre supplements or any use of probiotics in 2 months prior enrolment
* Unwillingness to exclude other probiotic products from diet during the study period

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-02-12 (Actual); Study Completion 2021-02-12 (Actual)

PRIMARY OUTCOMES:
Stool sample comparison | 56 days
  Comparison between samples at different taxonomical levels (phylum, family, genus and species) will be performed for the identification of specific bacteria in samples of interest. Accumulative bar charts will be provided for rapid inspection. PCA and clustering will be conducted. Biodiversity Index (Shannon, Simpson, Gini-Simpson or Berger-Parker) will be calculated. Biostatistics will be done in order to detect biomarkers between timepoints of the study.

SECONDARY OUTCOMES:
Fasting breath samples | 56 days
  Mean change in fasted breath hydrogen and methane, will be determined from baseline to end of study. Mean fasted hydrogen and mean fasted methane will be calculated independently of one each other. Breath hydrogen and breath methane will be measured in units of parts per million (ppm). Statistical significance will be determined using a paired t-test (p<0.05).
Bowel habit | 56 days
  Mean difference in stool frequency and consistency from baseline and end of study will be determined using a paired t-test, to determine significance (p<0.05).

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Hobson, Principal Investigator — The Functional Gut Clinic
Locations (1):
- The Functional Gut Clinic, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No